CLINICAL TRIAL: NCT05050019
Title: DIABETES DEVICE DISRUPTION DUE TO HOSPITALIZATIONS AND RADIOLOGIC PROCEDURES
Brief Title: DM DEVICE DISRUPTION SURVEY
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 202106074
Record Dates: First submitted 2021-09-09; First posted 2021-09-20 (Actual); Last update posted 2021-09-20 (Actual); Status verified 2021-09

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Rationale: Continuous glucose monitoring (CGM) and insulin pump therapy (CSII) have increased in utilization in the treatment of both type 1 and type 2 diabetes mellitus. Both types of devices are worn externally, with either a catheter or filament introduced into the subcutaneous space. Removal of these devices interrupts glucose monitoring or insulin delivery or both, which may have an adverse impact on patients' glucose control. Few studies have investigated the logistical and technical challenges that patients face when their insulin pump device or continuous glucose monitor (CGM) is interrupted.

Intervention: We will conduct a patient survey which seeks to identify and quantify the number of times insulin pump therapy or continuous glucose monitor has been disrupted, for what reason, how it was resolved and whether diabetes care had been adversely affected.

Objective: To determine the frequency and intensity of adverse health outcomes resulting from mandatory removal of CGM on insulin pump devices in healthcare or other settings.

Study population: Patients treated at Washington University outpatient clinics or Barnes Jewish Hospital between August 1, 2021- December 1, 2021. The study will include outpatients with diabetes mellitus who routinely utilize either CGM or insulin pump therapy or both. The target number of patients for the study will be 600, equally distributed between inpatients and outpatients, and with at least 100 having type 1 diabetes.

Study methodology: After providing consent, patients will complete an electronic questionnaire. Demographic information and diabetes history will be extracted from the patients' medical records.

Study endpoints: We will determine the incidence of disruptions to insulin pump therapy or continuous glucose monitoring in patients with diabetes mellitus as a result of hospitalization or medical test over a 1 year time period. We will also determine adverse health outcomes that resulted from device disruptions.

ELIGIBILITY:
Inclusion criteria

Female and male patients 18 years or older who meet all of the following criteria:

* Patients treated at Washington University outpatient clinics or Barnes Jewish Hospital.
* Patients with type 1 or type 2 diabetes mellitus who utilize CGM and/or insulin pump therapy.
* Patients who were able to read English.

Exclusion Criteria

* Patients who have not used a relevant device in the past 30 days
* Patients unwilling to or unable to provide consent or complete the questionnaire.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated at Washington University outpatient clinics or Barnes Jewish Hospital between August 1, 2021- December 1, 2021. The study will include outpatients with diabetes mellitus who routinely utilize either CGM or insulin pump therapy or both. The target number of patients for the study will be 600, equally distributed between inpatients and outpatients, and with at least 100 having type 1 diabetes.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-10-01 (Estimated); Primary Completion 2022-01-01 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
the incidence of disruptions to insulin pump therapy or continuous glucose monitoring in patients with diabetes mellitus as a result of hospitalization or medical test | over a 1 year time period
  Survey Responses

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Cedeno, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University, Barnes Jewish Hospital, St Louis, Missouri, United States